CLINICAL TRIAL: NCT04279756
Title: Comparing the Effects of Mobilization With Movement (MWM), Self MWM, and Dynamic Stretching on Hip Internal Rotation)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Cathy Arnot, Clinical Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00089974
Record Dates: First submitted 2020-01-17; First posted 2020-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hip; Anomaly
Keywords: Hip mobilization on hip internal rotation
MeSH Terms: conditions — Congenital Abnormalities | interventions — Movement

STUDY DESIGN:
Intervention Model Description: A parallel design, also called a parallel group study, compares two or more treatments. Participants are randomly assigned to either group, treatments are administered, and then the results are compared.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The care provider (Cathy Arnot) was not blinded as she knew the groups of the participants. The Investigators and the Outcomes Assessors were blinded as they were not aware of the group each participant was placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mildly Impaired Group (Active Comparator): This group is with participants with mildly impaired hip internal range of motion, from 25-30 degrees.
  Interventions: Other: Hip Mobilization with Movement, Self-Mobilization with Movement, Dynamic Stretch
- Moderately Impaired Group (Active Comparator): This group is with participants with moderately impaired hip internal range of motion, from 20-24 degrees.
  Interventions: Other: Hip Mobilization with Movement, Self-Mobilization with Movement, Dynamic Stretch
- Severely Impaired Group (Active Comparator): This group is with participants with severely impaired hip internal range of motion, less than 20 degrees.
  Interventions: Other: Hip Mobilization with Movement, Self-Mobilization with Movement, Dynamic Stretch

INTERVENTIONS:
Other: Hip Mobilization with Movement, Self-Mobilization with Movement, Dynamic Stretch — Participants receive either a therapist performed mobilization with movement, a self-mobilization with movement, or a dynamic stretch.

SUMMARY:
This study is looking to address the effectiveness of three different intervention on hip range of motion. There will be a therapist performed mobilization group, a self mobilization group, and a dynamic stretching group. Participants will be recruited from the University of South Carolina and randomly assigned between the three groups to have equal distribution and limit any biases. Participants will come in on two different days in order to receive the intervention on the first and have hip range of motion measured on both days. The investigators will be assessing if there is any significant difference between the three groups.

DETAILED DESCRIPTION:
The goal of this study is to compare the efficacy of three clinical interventions intended to treat hip dysfunctions such as hip osteoarthritis. Physical therapists utilize mobilization with movement clinically to increase range of motion that has been limited by hip pathology. This study will compare mobilization with movement administered by a physical therapist, self-administered mobilization with movement, in which patients are instructed in the maneuver and then perform it at home, and dynamic stretching as instructed by a physical therapist. Efficacy will be judged through changes in hip internal rotation range of motion, a motion which is typically limited in patients with hip pathology.

The objectives of the study are to quantify the effects of two different modalities of hip mobilization with movement and dynamic stretching in terms of hip internal rotation increases, and to inform current physical therapy practice by filling gaps in the literature surrounding the therapeutic effects of hip mobilization with movement. This study is intended to better equip physical therapists to select the most appropriate evidence-based interventions, thereby increasing the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* <30 degrees hip internal rotation in at least 1 hip

Exclusion Criteria:

* Traumatic injury in last 6 months
* FAI
* fracture
* surgery within last 6 months
* positive FADDIR/FABER
* symptomatic OA
* RA
* Neurologic conditions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Degrees of change in hip internal range of motion measured using a bubble inclinometer | Baseline, immediately post-intervention, 24 hours after intervention
  Degrees of change in hip internal range of motion will be measured before and after the intervention as well as a 24 hour follow up measurement to determine the duration of the increased range of motion before returning to baseline. All measurements will be taken using a bubble inclinometer which measures range of motion of a joint in degrees from 0-360.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Arnot, DPT, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
All data collected will be analyzed and interpreted only by the investigators listed for University of South Carolina and also investigators from Wingate University as they are also participating in the data collection.

REFERENCES:
- [Background] Hughes PE, Hsu JC, Matava MJ. Hip Anatomy and Biomechanics in the Athlete. Sports Medicine and Arthroscopy Review. 2002;10(2):103-114. doi:10.1097/00132585-200210020-00002.
- [Background] Moore KL, Dalley AF, Agur AMR. Clinically oriented anatomy. Philadelphia: Wolters Kluwer/Lippincott Williams & Wilkins Health; 2014.
- [Background] Byrne DP, Mulhall KJ, Baker JF. Anatomy & Biomechanics of the Hip. The Open Sports Medicine Journal. 2010;4(1):51-57. doi:10.2174/1874387001004010051.
- [Background] Simoneau GG, Hoenig KJ, Lepley JE, Papanek PE. Influence of hip position and gender on active hip internal and external rotation. J Orthop Sports Phys Ther. 1998 Sep;28(3):158-64. doi: 10.2519/jospt.1998.28.3.158. PMID 9742472
- [Background] Walsh R, Kinsella S. The effects of caudal mobilisation with movement (MWM) and caudal self-mobilisation with movement (SMWM) in relation to restricted internal rotation in the hip: A randomised control pilot study. Man Ther. 2016 Apr;22:9-15. doi: 10.1016/j.math.2016.01.007. Epub 2016 Jan 28. PMID 26995777
- [Background] Sadeghisani M, Manshadi FD, Kalantari KK, Rahimi A, Namnik N, Karimi MT, Oskouei AE. Correlation between Hip Rotation Range-of-Motion Impairment and Low Back Pain. A Literature Review. Ortop Traumatol Rehabil. 2015 Oct;17(5):455-62. doi: 10.5604/15093492.1186813. PMID 26751745
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Van Dillen LR, Bloom NJ, Gombatto SP, Susco TM. Hip rotation range of motion in people with and without low back pain who participate in rotation-related sports. Phys Ther Sport. 2008 May;9(2):72-81. doi: 10.1016/j.ptsp.2008.01.002. PMID 19081817
- [Background] Almeida GP, de Souza VL, Sano SS, Saccol MF, Cohen M. Comparison of hip rotation range of motion in judo athletes with and without history of low back pain. Man Ther. 2012 Jun;17(3):231-5. doi: 10.1016/j.math.2012.01.004. Epub 2012 Jan 26. PMID 22281524
- [Background] Albertin ES, Miley EN, May J, Baker RT, Reordan D. The Effects of Hip Mobilizations on Patient Outcomes: A Critically Appraised Topic. J Sport Rehabil. 2019 May 1;28(4):390-394. doi: 10.1123/jsr.2016-0238. Epub 2018 Dec 17. PMID 29466073
- [Background] Steultjens MP, Dekker J, van Baar ME, Oostendorp RA, Bijlsma JW. Range of joint motion and disability in patients with osteoarthritis of the knee or hip. Rheumatology (Oxford). 2000 Sep;39(9):955-61. doi: 10.1093/rheumatology/39.9.955. PMID 10986299
- [Background] Dekker J, Boot B, van der Woude LH, Bijlsma JW. Pain and disability in osteoarthritis: a review of biobehavioral mechanisms. J Behav Med. 1992 Apr;15(2):189-214. doi: 10.1007/BF00848325. PMID 1533877
- [Background] Shakoor N, Lee KJ, Fogg LF, Block JA. Generalized vibratory deficits in osteoarthritis of the hip. Arthritis Rheum. 2008 Sep 15;59(9):1237-40. doi: 10.1002/art.24004. PMID 18759259
- [Background] Bennell KL, Hinman RS. A review of the clinical evidence for exercise in osteoarthritis of the hip and knee. J Sci Med Sport. 2011 Jan;14(1):4-9. doi: 10.1016/j.jsams.2010.08.002. Epub 2010 Sep 17. PMID 20851051
- [Background] Beselga C, Neto F, Alburquerque-Sendin F, Hall T, Oliveira-Campelo N. Immediate effects of hip mobilization with movement in patients with hip osteoarthritis: A randomised controlled trial. Man Ther. 2016 Apr;22:80-5. doi: 10.1016/j.math.2015.10.007. Epub 2015 Oct 31. PMID 26559319
- [Background] Mulligan, B. R. (1993). Mobilisations with movement (MWM'S). Journal of Manual & Manipulative Therapy, 1(4), 154-156.
- [Background] Hsieh CY, Vicenzino B, Yang CH, Hu MH, Yang C. Mulligan's mobilization with movement for the thumb: a single case report using magnetic resonance imaging to evaluate the positional fault hypothesis. Man Ther. 2002 Feb;7(1):44-9. doi: 10.1054/math.2001.0434. No abstract available. PMID 11884156
- [Background] Kavanagh J. Is there a positional fault at the inferior tibiofibular joint in patients with acute or chronic ankle sprains compared to normals? Man Ther. 1999 Feb;4(1):19-24. doi: 10.1016/s1356-689x(99)80005-8. PMID 10463017
- [Background] Vicenzino B, Paungmali A, Teys P. Mulligan's mobilization-with-movement, positional faults and pain relief: current concepts from a critical review of literature. Man Ther. 2007 May;12(2):98-108. doi: 10.1016/j.math.2006.07.012. Epub 2006 Sep 7. PMID 16959529
- [Background] Yildirim MS, Ozyurek S, Tosun O, Uzer S, Gelecek N. Comparison of effects of static, proprioceptive neuromuscular facilitation and Mulligan stretching on hip flexion range of motion: a randomized controlled trial. Biol Sport. 2016 Mar;33(1):89-94. doi: 10.5604/20831862.1194126. Epub 2016 Feb 8. PMID 26929476
- [Background] Boykin RE, Stull JD, Giphart JE, Wijdicks CA, Philippon MJ. Femoroacetabular impingement in a professional soccer player. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1203-11. doi: 10.1007/s00167-012-2097-0. Epub 2012 Jul 3. PMID 22751941
- [Background] Burns SA, Mintken PE, Austin GP, Cleland J. Short-term response of hip mobilizations and exercise in individuals with chronic low back pain: a case series. J Man Manip Ther. 2011 May;19(2):100-7. doi: 10.1179/2042618610Y.0000000007. PMID 22547920
- [Background] Abbott JH. Mobilization with movement applied to the elbow affects shoulder range of movement in subjects with lateral epicondylalgia. Man Ther. 2001 Aug;6(3):170-7. doi: 10.1054/math.2001.0407. PMID 11527457
- [Background] Vicenzino B, Branjerdporn M, Teys P, Jordan K. Initial changes in posterior talar glide and dorsiflexion of the ankle after mobilization with movement in individuals with recurrent ankle sprain. J Orthop Sports Phys Ther. 2006 Jul;36(7):464-71. doi: 10.2519/jospt.2006.2265. PMID 16881463
- [Background] Bandy WD, Irion JM, Briggler M. The effect of static stretch and dynamic range of motion training on the flexibility of the hamstring muscles. J Orthop Sports Phys Ther. 1998 Apr;27(4):295-300. doi: 10.2519/jospt.1998.27.4.295. PMID 9549713
- [Background] Lachtman DS, Bartha DA, Beltran MM, Dominguez DN, Messerli AR, Miller SE, Davis AM, Nelson-Wong E. Rater Reliability and Concurrent Validity of Single and Dual Bubble Inclinometry to Assess Cervical Lateral Flexion. J Manipulative Physiol Ther. 2015 Oct;38(8):572-80. doi: 10.1016/j.jmpt.2015.08.003. Epub 2015 Sep 26. PMID 26391235
- [Background] Kolber MJ, Pizzini M, Robinson A, Yanez D, Hanney WJ. The reliability and concurrent validity of measurements used to quantify lumbar spine mobility: an analysis of an iphone(R) application and gravity based inclinometry. Int J Sports Phys Ther. 2013 Apr;8(2):129-37. PMID 23593551

DOCUMENTS (2):
  • Study Protocol (2020-02-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT04279756/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT04279756/SAP_001.pdf